CLINICAL TRIAL: NCT04311905
Title: Efficiency of Diode Laser Activated Irrigation on Healing of Periapical Tissues (A Randomized Clinical Trial )
Brief Title: Efficiency of Diode Laser Activated Irrigation on Healing of Periapical Tissues
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Hend Hamdy Ismail, PhD candidate, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: END 16-15D
Record Dates: First submitted 2020-03-07; First posted 2020-03-17 (Actual); Last update posted 2020-03-18 (Actual); Status verified 2020-03

CONDITIONS: Periapical Diseases
Keywords: Diode laser; CBCT; low level laser therapy
MeSH Terms: conditions — Periapical Diseases | interventions — Lasers, Semiconductor

STUDY DESIGN:
Who Masked: Participant
Masking Description: Single blinded
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Laser activated irrigation LAI (Experimental): Diode Laser activated irrigation
  Interventions: Device: Diode laser
- conventional root canal treatment (Placebo Comparator): mock LAI , conventional root canal treatment 2.5% sodium hypochlorite
  Interventions: Other: Placebo

INTERVENTIONS:
Device: Diode laser — Diode laser activated irrigation
  Other Names: LAI
  Arms: Laser activated irrigation LAI
Other: Placebo — mock Laser activated irrigation
  Arms: conventional root canal treatment

SUMMARY:
Study is a Randomized clinical trial conducted at Endodontic department- Ain Shams university Cairo. Egypt. 24 eligible patients were selected and included in the study to compare healing ability of diode laser activated irrigation versus conventional root canal treatment using CBCT

DETAILED DESCRIPTION:
Sample size is 24 , 24 Patients were randomly distributed in 2 groups , one group of patients received laser activated irrigation LAI during root canal treatment and the other group received no treatment just conventional RCT. • Patients were equally divided into 2 groups (n=12 in each group ) The study in a Single blinded RCT , Numbers for patients will be generated and distributed randomly in a table on an Excel sheet, and in front of each number either a letter (C) for control or (I) for intervention will be typed After patients were selected in the study they will be asked to fill in a consent form , that states that they are part of a clinical trial and that they may or may not receive a laser activated irrigation Group A LAI :Disinfection were done by using 5 ml of 2.5% sodium hypochlorite irrigation for 1 minute. Irrigation will be performed with a 30-gauge needle side vented The irrigation needles were introduced passively up to 2 mm away the working length. After irrigation Laser treatment will be performed with a diode laser, at a wavelength of 980 nm with a repeated pulse mode using a pulse duration of 5sec per canal and a pulse interval of 0.2 ms. The laser irradiation were delivered for 1 minute into the canal up to 1 mm short of the working length, with circling movements from the apical part moving towards the coronal part Group B : received mock laser intervention , conventional Root canal treatment with 2.5% sodium hypochlorite CBCT was taken pre-operative and another one was taken after 12 month , both volumetric and linear measurements were calculated

ELIGIBILITY:
Inclusion Criteria:

* Adult patients age between 18-50 years
* Medically free patients.
* Patients suffering from acute or chronic infection with symptomatic apical periodontitis with Necrotic pulp
* Preoperative Pain
* Sensitivity to percussion
* Periapical radiographic X-ray showing periapical lesion with no gutta percha in canal
* Occlusal contact with opposing teeth

Exclusion Criteria:

* Pregnant females.
* Patients having a significant systemic disorder or history of drug abuse
* Patients who had administrated analgesics or antibiotics during the last 12 hours preoperatively.
* Patients having bruxism or clenching
* Teeth having:

  * No occlusal contact
  * No sensitivity to percussion
  * Greater than grade I mobility.
  * Pocket depth greater than 5mm.
  * No possible restorability
  * Procedural errors
  * Previous Root canal treatment
  * Open apex

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2017-07-01 (Actual); Primary Completion 2019-07-01 (Actual); Study Completion 2020-01-01 (Actual)

PRIMARY OUTCOMES:
Assess post-operative healing using CBCT in a period of 12 month when Laser activated irrigation was used during root canal treatment | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Maram Obeid, PhD, Study Director — AinShams University; Ehab Hassanien, PhD, Study Chair — Ainshams University
Locations (1):
- Endodontic department - Faculty of Dentistry Ainshams University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hamdy Ismail H, Obeid MF, ElSaid Hassanein E. The efficiency of single-session photobiomodulation on healing of periapical bone lesions using CBCT: a randomized clinical trial. Lasers Med Sci. 2025 Jan 23;40(1):31. doi: 10.1007/s10103-024-04242-5. PMID 39847087